CLINICAL TRIAL: NCT01092897
Title: Biomarkers in Pulmonary Arterial Hypertension Treated With Imatinib
Brief Title: Pulmonary Hypertension and Imatinib
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kewal Asosingh, Ph.D, Associate Staff, The Cleveland Clinic
Other Study IDs: 09-782
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: PAH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with PAH treated with Imatinib

SUMMARY:
The purpose of the study is to determine whether circulating molecular and cellular biomarkers are predictive of imatinib effect on pulmonary artery hypertension.

DETAILED DESCRIPTION:
We hypothesize that bone marrow progenitor cells are mobilized into the circulation in PAH, home to the lungs and differentiate into mast cells, which promote vascular remodeling and vasoconstriction through release of renin and chymase. As a corollary to this, we hypothesize that anti cKit tyrosine kinase inhibitor (TKI), imatinib, provides clinical benefit to patients through inhibition of mast cell progenitor proliferation, mobilization and differentiation. To test this, we will determine if mast cell progenitors and mast cell biomarkers are related to imatinib clinical response. This will be an ancillary study, part of a placebo-controlled, double-blind multi center clinical trial of imatinib in pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

from Imatinib Trial

* Male or Female 18 years or older
* A current diagnosis or Pulmonary Arterial Hypertension according to the Dana Point 2008 Meeting: WHO Diagnostic Group I, idiopathic or heritable (familial or sporadic) PAH, PAH associated with collagen vascular disease including systemic sclerosis, rheumatoid arthritis, mixed connective tissue diseases, and overlap syndrome. PAH following one year repair of congenital heart defect (ASD, VSD, or PDA), or PAH associated with diet therapies or other drugs
* A PVR>1000dynes.sec.cm-5(as assess by RHC at screening or in the 2 months preceding the screening visit despite treatment with two or more specific PAH therapies, including endothelin receptor antagonists (ERA), phosphodiesterase 5 inhibitors (PDE5), or inhaled, intravenous or oral prostacyclin analogues for ≥3 months. On stable background therapy doses for ≥ 30 days except for warfarin (≥30 days but doses can vary even within the mouth before enrollment)
* WHO Functional Class II-IV. For WHO Functional Class IV, one of the 2 or more specific PAH therapies must be an inhaled, intravenous or oral prostacyclin analogue, unless the subject has been shown to be intolerant of prostacyclin analogues.
* 6MWD≥150meters and ≥450meters at screening. Distances of two consecutive 6MWTs should be within 15% of one another.
* Ability to provide written informed consent

Exclusion Criteria: from Imatinib Trial

* Women of childbearing potential who are not practicing birth control methods.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of positive hCG laboratory test (> 5 mIU/MI)
* Have previously received treatment with imatinib
* In treatment with chronic nitric oxide therapy
* Pre-existing lung disease including parasitic diseases affecting lungs, congenital abnormalities of the lungs, thorax or diaphragm or bronchial asthma associated with chronic hypoxia that may contribute to severity of PAH
* With a pulmonary capillary wedge pressure >15 mm Hg to rule out PAH secondary to left ventricular dysfunction
* With a diagnosis of pulmonary artery or vein stenosis
* With other diagnosis of PAH in WHO Diagnostic Group 1 re excluded including congenital systemic to pulmonary shunts (large, small that not surgically repaired, portal hypertension, HIV infection, glycogen storage disease, Gaucher's disease, hereditary hemorrhagic telangiectasia, hemoglobinopthaies, myeloproliferative disorders)
* With a diagnosis of PAH associated with: venous hypertension (WHO Diagnostic Group II), hypoxia (WHO Diagnostic Group III), chronic pulmonary thromboembolic disease (WHO Diagnostic Group IV) or other miscellaneous causes (WHO Diagnostic Class V, which includes sarcoidosis, histiocytosis X, lympangiomatosis, compression of pulmonary vessels).
* With deficient thrombocyte function, thrombocytopenia >50x109/L(50x103/µL)
* With a history of acute heart failure or chronic left sided heart failure
* With uncontrolled systemic arterial hypertension, systolic >160mmHg or diastolic >90mmHg
* With hemoglobin <100g/L (10 g/dl)
* With deficiencies of blood coagulation, inherited or acquired blood disorders, factor XII, factor XIII; decreased generation of coagulation factors due to acute or chronic liver diseases, efficient coagulation due to auto-antibodies against coagulation factors such as in lupus anticoagulant
* With disseminated intravascular coagulation (DIC)
* With evidence of major bleeding or intracranial hemorrhage
* With a history of latent bleeding risk such as diabetic retinopathy, gastrointestinal bleeding due to gastric or duodenal ulcers, or colitis ulcerosa
* With a history of moderate or greater hepatic insufficiency transaminase levels >4times the upper limit or normal or a bilirubin >2times the upper limit of normal
* With a history of renal insufficiency (serum creatinine >200µmol/1or 2.6mg/dl)
* Previous therapeutic radiation of lungs mediastinum
* With a history of sickle cell anemia
* With a QTcF>450msec for males and >470 msec for females at screening
* With a history of ventricular tachycardia, ventricular fibrillation or ventricular flutter
* Having syncope in the 3 months prior to the screening visit
* With a history of Torsades de Pointes
* With a history of long QT syndrome
* Having undergone atrial septostomy in the 3 months prior to screening visit
* Having undergone radiofrequency catheter ablation for atrial or sinus arrhythmias in the 3 months prior to screening visit
* With an advanced, sever, or unstable disease of any type that may interfere with the primary and secondary endpoint evaluations
* With a history of immunodeficiency diseases, including HIV
* With a known hypersensitivity to QTI571 or drugs similar to the study drug
* With a disability that may prevent the patient from competing all study requirements and in particular, interfere with the 6MWT assessment
* With a life expectancy of 6months or less
* Having used other investigational drugs at the time of enrollment, within 30 days or 5 half-lives of enrollment, whichever is longer
* With a history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* With a diagnosis of Hepatitis B or C
* With a history of alcohol abuse within 6 months of screening
* With a history of illicit drug abuse within 6 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with PAH that are enrolled in the Imatinib clinical trial.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measuring circulating biomarkers of imatinib affect | within one year of the end of the study

SECONDARY OUTCOMES:
Evaluate effect of imatinib on the activation of mast cells | within one year of the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Kewal Asosingh, M.S., Ph.D, Principal Investigator — The Cleveland Clinic
Locations (8):
- United States (8):
  - University of Colorado Denver, Aurora, Colorado
  - Cleveland Clinic Florida, Weston, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center of Dallas, Dallas, Texas

REFERENCES:
- [Background] Patterson KC, Weissmann A, Ahmadi T, Farber HW. Imatinib mesylate in the treatment of refractory idiopathic pulmonary arterial hypertension. Ann Intern Med. 2006 Jul 18;145(2):152-3. doi: 10.7326/0003-4819-145-2-200607180-00020. No abstract available. PMID 16847299
- [Background] Schermuly RT, Dony E, Ghofrani HA, Pullamsetti S, Savai R, Roth M, Sydykov A, Lai YJ, Weissmann N, Seeger W, Grimminger F. Reversal of experimental pulmonary hypertension by PDGF inhibition. J Clin Invest. 2005 Oct;115(10):2811-21. doi: 10.1172/JCI24838. PMID 16200212
- [Background] Dentelli P, Rosso A, Balsamo A, Colmenares Benedetto S, Zeoli A, Pegoraro M, Camussi G, Pegoraro L, Brizzi MF. C-KIT, by interacting with the membrane-bound ligand, recruits endothelial progenitor cells to inflamed endothelium. Blood. 2007 May 15;109(10):4264-71. doi: 10.1182/blood-2006-06-029603. Epub 2007 Feb 8. PMID 17289809
- [Background] Heath D, Yacoub M. Lung mast cells in plexogenic pulmonary arteriopathy. J Clin Pathol. 1991 Dec;44(12):1003-6. doi: 10.1136/jcp.44.12.1003. PMID 1791199
- [Background] Hamada H, Terai M, Kimura H, Hirano K, Oana S, Niimi H. Increased expression of mast cell chymase in the lungs of patients with congenital heart disease associated with early pulmonary vascular disease. Am J Respir Crit Care Med. 1999 Oct;160(4):1303-8. doi: 10.1164/ajrccm.160.4.9810058. PMID 10508822